CLINICAL TRIAL: NCT03568578
Title: A Study in Reversing Hepatic Fibrosis or Cirrhosis Related to Hepatitis B Virus and Finding Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Principal Investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017ZX10203202002
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B; Liver Fibrosis
Keywords: Fibrosis; Liver Cirrhosis; non-invasive biopsy; hepatitis B virus
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Fibrosis | interventions — entecavir; anluohuaxian

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir Group (Active Comparator): Patients in this arm will be given Entecavir 0.5 mg a day for 2 years.
  Interventions: Drug: Entecavir 0.5 mg
- Entecavir and Anluohuaxian Group (Experimental): Patients in this arm will be given Entecavir 0.5 mg and Anluohuaxian Pill 12 g a day for 2 years.
  Interventions: Drug: Entecavir 0.5 mg; Drug: Anluohuaxian Pill 12g

INTERVENTIONS:
Drug: Entecavir 0.5 mg — Patients in this group will be given Entecavir 0.5 mg a day for 2 years.
  Other Names: ETV
Drug: Anluohuaxian Pill 12g — Patients in this group will be given Entecavir 0.5 mg and Anluohuaxian Pill 12g a day for 2 years
  Other Names: ALHX
  Arms: Entecavir and Anluohuaxian Group

SUMMARY:
The aim of our study is to validate the non-invasive model which was constructed by our previous study for evaluating liver fibrosis or cirrhosis caused by hepatitis B virus in mainland China and to find a therapeutic regimen to reverse liver fibrosis and cirrhosis.

DETAILED DESCRIPTION:
450 patients who are infected with hepatitis B virus for at least 6 months will be included in the study. They will be divided into two groups. One group will be treated with Entecavir while another treated with Entecavir and Anluohuaxian Pill. Liver biopsy samples and blood samples from the patients will be used to validate the non-invasive model. Furthermore, the samples will be used to evaluate if Anluohuaxian Pill could reverse liver fibrosis and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg positive for at least 6 months
2. Agree to have liver biopsy
3. Male or female aged 18 to 70 years old -

Exclusion Criteria:

1. Patients with alcoholic liver disease, autoimmune liver disease, heretic liver disease, drug induced liver disease, nonalcoholic liver disease or other chronic liver disease
2. Platelet count < 80 × 10^9/L
3. Prothrombin activity ≤ 60%
4. Decompensated liver cirrhosis
5. Patients with any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Construct a non-invasive model based on laboratory tests | 26 weeks after liver biopsy
  We will measure the following biomarkers: TIMP1，CXCL10，CD25，YKL-40，collagen IV，von Willebrand Factor，TGF-β1，ANGPTL2，MMP-9，IL-2R，PDGF-AA，PDGF-BB，TGF-a，LN，MMP-1, soluble CD163 and CXCL9. To formulate the predictive models for detecting significant fibrosis (Ishak fibrosis score ≥3)， univariate analysis was performed on variables between patients with and without significant fibrosis. The significant variables (p<0.05) were then subjected to multivariate stepwise logistic regression, using backward approaches, and were combined using the logistic regression function. The diagnostic value of each regression model was assessed using receiver operating characteristics curves.

SECONDARY OUTCOMES:
Compare the difference of fibrosis reverse rates between the two groups | 26 weeks after liver biopsy
  Liver biopsy samples will be evaluated by Ishak fibrosis score. Then we compare the difference of fibrosis reverse rates between the two groups by Ishak fibrosis score.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (16):
- China (16):
  - Guiqiang Wang, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi the Fifth People's Hospital, Wuxi, Jiangsu
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang First Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Li J, Dong XQ, Cao LH, Zhang ZQ, Zhao WF, Shang QH, Zhang DZ, Ma AL, Xie Q, Gui HL, Zhang G, Liu YX, Shang J, Xie SB, Liu YQ, Zhang C, Wang GQ, Zhao H; China HepB Related Fibrosis Assessment Research Group. Factors associated with persistent positive in HBV DNA level in patients with chronic Hepatitis B receiving entecavir treatment. Front Cell Infect Microbiol. 2023 Jun 16;13:1151899. doi: 10.3389/fcimb.2023.1151899. eCollection 2023. PMID 37396307